CLINICAL TRIAL: NCT05343988
Title: Percutaneous Neurostimulation for Treatment of Paroxysmal Sympathetic Hyperactivity in Children With Acute Severe Brain Injury
Brief Title: Percutaneous Neurostimulation to Treat Paroxysmal Sympathetic Hyperactivity in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Binod Balakrishnan, MD, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1817951
Record Dates: First submitted 2022-04-10; First posted 2022-04-25 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Paroxysmal Sympathetic Hyperactivity
Keywords: peripheral neurostimulator; pediatric; acute severe brain injury

STUDY DESIGN:
Intervention Model Description: Prospective unblinded pilot study to evaluate the feasibility of use of a peripheral neurostimulator for treatment of paroxysmal sympathetic hyperactivity in children with acute severe brain injury
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Percutaneous Electrical Nerve Field Stimulation (PENFS) device application (Experimental): The peripheral neurostimulator, PENFS device, will be placed over the external ear of enrolled patients. The device will continuously stay in place for 120 hours.
  Interventions: Device: Percutaneous Electrical Nerve Field Stimulation (PENFS) device application

INTERVENTIONS:
Device: Percutaneous Electrical Nerve Field Stimulation (PENFS) device application — PENFS device will be used to treat children with paroxysmal sympathetic hyperactivity (PSH) due to acute severe brain injury.
  Other Names: Peripheral neurostimulator

SUMMARY:
Survivors of severe brain injury, such as lack of oxygen or severe traumatic brain injury, frequently experience Paroxysmal Sympathetic Hyperactivity (PSH). PSH is characterized by disabling symptoms such as a fast heart rate, high blood pressure, rapid breathing, rigidity, tremors, and sweating due to uncontrolled sympathetic hyperactivity in the nervous system. Effective treatment is necessary to decrease secondary brain injury, prevent weight loss from increased metabolic demand and reduce suffering. Currently, a combination of medications to slow down the sympathetic nervous system, muscle relaxants, anti-anxiety drugs, gabapentin, and narcotics are used to treat PSH. The sudden, recurrent attacks of PSH often require repeated rescue medications and multiple drugs with a high risk of side effects. Non-drug treatments for PSH may revolutionize treatment. The novel and non-invasive Percutaneous Electrical Nerve Field Stimulation (PENFS) device is an attractive and potentially effective treatment option for PSH.

PENFS, applied to the external ear, has been shown to be effective for conditions such as abdominal pain, narcotic withdrawal, and cyclic vomiting syndrome, all which have similar symptoms to PSH. Therefore, the hypothesis is PENFS could be effective in the treatment of PSH. The electrical current delivered by the PENFS device is thought to increase parasympathetic activity by stimulating a branch of the vagus nerve. PENFS was shown to decrease central sympathetic nervous system activity by 36% within 5 minutes of being placed in the ear of a rat model. Similar central inhibition could improve symptoms of PSH. This pilot study aims to evaluate the feasibility of performing an efficacy trial of PENFS for children with PSH.

DETAILED DESCRIPTION:
Paroxysmal sympathetic hyperactivity - incidence, pathophysiology, diagnosis, treatment, prognosis and implications for treatment Paroxysmal sympathetic hyperactivity is frequently seen in survivors of acute severe brain injury (ASBI). It is most commonly associated with severe traumatic brain injury (sTBI) with a reported incidence of 10-20% among survivors of sTBI. Survivors of anoxic brain injury have a higher incidence of PSH (approximately 30%). The pathophysiology of PSH is incompletely understood. Current consensus is that it the result of disconnection between with neuroinhibitory higher centers in the diencephalon and the excitatory pathways in the brainstem and spinal cord (10). PSH is characterized by a constellation of symptoms such as tachycardia, tachypnea, hypertension, hyperthermia, rigidity, tremors, sweating, and pupillary dilation as a result of sympathetic hyperactivity due to the brain injury. Research on PSH has been hampered by lack of a uniform definition and use of various terms such as neurostorming, dysautonomia. Consensus diagnostic criteria and a scoring algorithm (CFS) were developed in 2014 (Table 1a,1b). This tool has 2 components - Clinical Feature Scale to score the severity of symptoms and Diagnosis Likelihood Tool (DLT) that lists the diagnostic features to help with initial diagnosis of PSH (Table 1b). The combined CFS and DLT scores are used to assess the likelihood of PSH (Table 1b). We will use a CFS+DLT cut-off of ≥ 10 to diagnose PSH. PSH increases the risk for secondary brain injury and is associated with worse functional outcomes, longer hospitalization and higher healthcare costs. Appropriate treatment of PSH is important for patient comfort and to prevent secondary brain damage.

Currently, PSH is treated using a combination of multiple neurotropic medications (narcotics, benzodiazepines, sympatholytics, gabapentin, muscle relaxants etc.) that can result in complications due to their side effects such as excessive sedation, respiratory depression, drug dependence, and constipation. Some of these medications necessitate ICU stay due to their CNS depressant effects thus potentially increasing healthcare costs. There has been very little research into novel ways of treating PSH other than the use of various neurotropic medications.

Measurement of autonomic function - HRV and Pupillometry Autonomic function can be evaluated clinically and is most commonly measured using heart rate variability (HRV). Established standards for measurement of HRV are available. HRV has been studied in various disease states in the intensive care environment such as post-acute MI, sepsis, multi-organ dysfunction, brain injury, and brain death. HRV is decreased or lost in severe disease and has been shown to be associated with increased mortality in the ICU. Higher sympathetic activity in severe disease states is associated with decreased HRV. HRV was shown to be significantly different between children and adults with ASBI and controls. Similarly, pupillary reactivity is also under autonomic control. Recently, pupillometry has also been used to measure autonomic activity. A pupillometer quantitatively measures pupil size (size, minimum size with light stimulus, % change in pupil size) and reactivity (constriction velocity, max constriction velocity, latency, dilation velocity) that can be compared to established norms and trended over time. These parameters have been shown to reflect sympathetic (dilation velocity) and parasympathetic system (% change in pupil size, latency, constriction velocity) activity and sympatho-parasympathetic balance (baseline pupil size). PSH, as the name implies, is associated with uncontrolled paroxysms of sympathetic activity that results in pupillary dilation among other symptoms. It is conceivable that an increase in parasympathetic activity would alter these parameters that could be compared using the patient as his/her own control.

PENFS device - description, mechanism of action, and applications The PENFS (auricular neurostimulator) device is a novel, non-pharmacological therapy that has been effectively used for various conditions such as functional abdominal pain, chronic pain, and narcotic withdrawal. Recent data from CW also demonstrates efficacy in a pilot study for children with cyclic vomiting syndrome, with improvement in episode severity and frequency lasting an average 5 months (unpublished data). Cyclic vomiting syndrome (CVS) is a disorder of autonomic imbalance manifested by severe sympathetic hyperactivity. Symptoms of nausea/vomiting, pallor, diaphoresis, and tachycardia are similar to PSH. Many of the symptoms of narcotic withdrawal are also very similar to those of PSH including tachycardia, tachypnea, hypertension, fever, tremors, and sweating. Clonidine, an alpha-2 agonist with sympatholytic properties is commonly used as an adjunct in the treatment of narcotic withdrawal syndrome. Clonidine is also one of the first-line medications used for treatment of PSH. Thus, it is plausible that PENFS could be effective in treatment of PSH.

The PENFS device is applied over the external ear and is continuously worn for 120 hours at a time. The electrical current stimulates the auricular branch of the vagus nerve (ABVN) and auricular branches of cranial nerves V, VII and IX. The nerves project to the various parts of the brain, including the brainstem nucleus tractus solitarius. fMRI scans in healthy human volunteers have shown significant activation of the central vagal projections by stimulating ABVN. Sympathoinhibition has been shown to be one of the primary mechanisms of action of the device in the various conditions for which it is used. Electrical stimulation of the tragus has been shown to cause central sympathoinhibition in rats by up to 36% within 5 minutes of stimulation. This central sympathoinhibition by the PENFS device could improve the symptoms of PSH.

One of the advantages of PENFS in the treatment of PSH is that it is continuously active while it is worn thus providing symptomatic treatment throughout that period. This could help prevent or ameliorate the paroxysmal symptoms classically seen in PSH and thus reduce the need for rescue medications. The device also has been shown to have a relatively rapid onset of action. A recent study showed that the onset of action was rapid with 63% reduction in narcotic withdrawal score within 20 minutes of activation of the device and 85% reduction within 60 minutes. Thus, PENFS could offer a non-pharmacological tool for managing PSH, helping to decrease the need for maintenance and rescue medications and thus limiting the side effects of some of these medications. Decreased need for neurosedative medications could further decrease the length of ICU stay for these patients thus decreasing healthcare costs. The device is also well-tolerated without any serious adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-17 years age with PSH due to ASBI
* PSH severity score > 6 (moderate severity)
* Glasgow Coma Scale < 15

Exclusion Criteria:

* age < 2 years (small ears thus less surface area to apply the leads)
* ear deformity or severe dermatitis of ear lobes,
* intractable seizures, heart block, patients with other implantable devices (cardiac pacemaker, vagal nerve stimulator, etc.
* known pregnancy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The number of children enrolled (Ages 2-17) with acute severe brain injury (ASBI) and Paroxysmal Sympathetic Hyperactivity (PSH) to use the Percutaneous Electrical Nerve Field Stimulation (PENFS) device for treatment | Up to 192 hours.
  Number of patients enrolled
Study retention for those children enrolled with acute severe brain injury (ASBI) and Paroxysmal Sympathetic Hyperactivity (PSH) to use the Percutaneous Electrical Nerve Field Stimulation (PENFS) device for treatment | Up to 192 hours.
  Percentage of patients who complete the study
Device tolerability for those children enrolled with acute severe brain injury (ASBI) and Paroxysmal Sympathetic Hyperactivity (PSH) to use the Percutaneous Electrical Nerve Field Stimulation (PENFS) device for treatment | Up to 192 hours.
  Percentage of patients withdrawn due to device intolerability
Capturing at least 80 percent of scoring events to assess pediatric Paroxysmal Sympathetic Hyperactivity (PSH) symptoms using the Clinical Feature Severity (CFS) scoring tool | Up to 192 hours.
  The CFS will be administered by trained bedside nurses to capture PSH severity in enrolled patients before, during and after initiation of PENFS device treatment. The CFS is a composite measure of Heart Rate, Respiratory Rate, Systolic Blood Pressure, Temperature, Sweating and Posturing. The Scoring is as follows: 0 Nil; 1-6 Mild; 7-12 Moderate; and >=13 Severe. Percentage of CFS scores collected.

SECONDARY OUTCOMES:
The change from baseline of the Clinical Feature Scale (CFS) measured throughout the study to 192 hours after device placement | 0 hours before device placement, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 84 hours, 96 hours, 108 hours,120 hours-device discontinuation, 132 hours, 144 hours, 156 hours, 168 hours, 180 hours, 192 hours
  The CFS is a composite measure of Heart Rate, Respiratory Rate, Systolic Blood Pressure, Temperature, Sweating and Posturing designed to measure the severity of Paroxysmal Sympathetic Hyperactivity (PSH). The Scoring of PSH is as follows: 0 Nil; 1-6 Mild; 7-12 Moderate; and >=13 Severe. The before and after (192hrs) will be analyzed along with the trend in score over time.
Measure a change in maintenance and rescue medication use for treatment of PSH | 0-24hours, 25-48hours, 49-72hours, 73-96hours, 97-120hours
  Maintenance medications and the number of doses and type of rescue medications administered will be collected for enrolled patients every 24 hours. These will be compared to a historical cohort of PSH patients (2-17 years old) identified using the ICU Neurology database from January 2018 - August 2021. The association of the CSF score and the number of doses of maintenance and rescue medications will be summarized with a spearman correlation coefficient and exact 95% Confidence intervals (CI).
Measure pupil size (mm) to determine the change in autonomic response | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by using pupillometry to measure pupil size during the 12-hour period before and after initiation of PENFS therapy. Pupillometry is standard of care for monitoring ASBI patients. Enrolled patients would have pupillometry readings available even prior to initiation of PENFS.
Measure pupil's constriction velocity (mm/sec) to determine the change in autonomic response | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The Percutaneous Electrical Nerve Field Stimulation (PENFS) device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by using pupillometry to measure the constriction velocity during the 12-hour period before and after initiation of PENFS therapy. Pupillometry is standard of care for monitoring ASBI patients. Enrolled patients would have pupillometry readings available even prior to initiation of PENFS.
Measure the pupil's dilation velocity (mm/sec) to determine the change in autonomic response | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The Percutaneous Electrical Nerve Field Stimulation (PENFS) device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by using pupillometry to measure the dilation velocity during the 12-hour period before and after initiation of PENFS therapy. Pupillometry is standard of care for monitoring ASBI patients. Enrolled patients would have pupillometry readings available even prior to initiation of PENFS.
Measure the change in Heart Rate Variability (HRV) parameter: Standard Deviation of NN Intervals (SDNN) (msec) to determine the change in autonomic response with Percutaneous Electrical Nerve Field Stimulation (PENFS) use | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The Percutaneous Electrical Nerve Field Stimulation (PENFS) device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by measuring SDNN as part of evaluation of HRV during the 12-hour period before and after initiation of PENFS therapy. Higher scores are better as evidenced by greater HRV.
Measure the change in the Heart Rate Variability (HRV) parameter: Root Mean Square of the Successive Differences (RMSSD) to determine the change in autonomic response with the Percutaneous Electrical Nerve Field Stimulation (PENFS) device use | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The Percutaneous Electrical Nerve Field Stimulation (PENFS) device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by measuring RMSSD as part of evaluation of HRV during the 12-hour period before and after initiation of PENFS therapy. Higher scores are better as evidenced by greater HRV.
Measure the change in the Heart Rate Variability (HRV) parameter: Total power (TP) (ms^2) to determine the change in autonomic response with Percutaneous Electrical Nerve Field Stimulation (PENFS) use | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The PENFS device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by measuring Total power (TP) as part of evaluation of HRV during the 12-hour period before and after initiation of PENFS therapy.
Measure the change in the Heart Rate Variability (HRV) parameter: High Frequency (HF) (ms^2) to determine the change in autonomic response with Percutaneous Electrical Nerve Field Stimulation (PENFS) use | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The PENFS device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by measuring High Frequency (HF) as part of evaluation of Heart Rate Variability (HRV) during the 12-hour period before and after initiation of PENFS therapy. Higher values are better.
Measure the change in the Heart Rate Variability (HRV) parameter Low frequency (LF) to determine the change in autonomic response with Percutaneous Electrical Nerve Field Stimulation (PENFS) use | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The PENFS device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by measuring Low Frequency (LF) (ms^2) as part of evaluation of HRV during the 12-hour period before and after initiation of PENFS therapy. Higher values are better.
Measure the change in the Heart Rate Variability (HRV) parameter: Low Frequency: High Frequency (LF:HF) ratio to determine the change in autonomic response with Percutaneous Electrical Nerve Field Stimulation (PENFS) use | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The PENFS device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by measuring LF:HF ratio as part of evaluation of HRV during the 12-hour period before and after initiation of PENFS therapy. A higher number indicates increased sympathetic activity or reduced parasympathetic activity.
Measure the change in the HRV parameter: Mean Heart Rate (Mean HR) (beats per minute/bpm) to determine the change in autonomic response with Percutaneous Electrical Nerve Field Stimulation (PENFS) use | -12 hours (12 hours before placement), Time 12 hours (12 hours after placement)
  The PENFS device will be tested to determine if it results in higher parasympathetic activity due to stimulation of the auricular branch of the vagus nerve. This will be assessed by measuring the change in (Mean HRT) Mean Heart Rate as part of evaluation of HRV during the 12-hour period before and after initiation of PENFS therapy. Normal HRT is between 60-90 beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Binod Balakrishnan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in the publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of results - for up to 3 years
Access Criteria: De-identified, individual participant data including a data dictionary will be made available through encrypted e-mail immediately after publication for 3 years. Researchers who provide a proposal, directed to jbergholte@mcw.edu, will be required to enter into a Data Use Agreement with the Medical College of Wisconsin and demonstrate in a written statement how the data relates to the proposal's objectives. In addition, the Study Protocol, Informed Consent, Statistical Analysis Plan and Clinical Study Report will be made available.

REFERENCES:
- [Background] Fernandez-Ortega JF, Prieto-Palomino MA, Munoz-Lopez A, Lebron-Gallardo M, Cabrera-Ortiz H, Quesada-Garcia G. Prognostic influence and computed tomography findings in dysautonomic crises after traumatic brain injury. J Trauma. 2006 Nov;61(5):1129-33. doi: 10.1097/01.ta.0000197634.83217.80. PMID 17099518
- [Background] Baguley IJ, Slewa-Younan S, Heriseanu RE, Nott MT, Mudaliar Y, Nayyar V. The incidence of dysautonomia and its relationship with autonomic arousal following traumatic brain injury. Brain Inj. 2007 Oct;21(11):1175-81. doi: 10.1080/02699050701687375. PMID 17952716
- [Background] Rabinstein AA. Paroxysmal sympathetic hyperactivity in the neurological intensive care unit. Neurol Res. 2007 Oct;29(7):680-2. doi: 10.1179/016164107X240071. PMID 18173907
- [Background] Kirk KA, Shoykhet M, Jeong JH, Tyler-Kabara EC, Henderson MJ, Bell MJ, Fink EL. Dysautonomia after pediatric brain injury. Dev Med Child Neurol. 2012 Aug;54(8):759-64. doi: 10.1111/j.1469-8749.2012.04322.x. Epub 2012 Jun 19. PMID 22712762
- [Background] Fernandez-Ortega JF, Prieto-Palomino MA, Garcia-Caballero M, Galeas-Lopez JL, Quesada-Garcia G, Baguley IJ. Paroxysmal sympathetic hyperactivity after traumatic brain injury: clinical and prognostic implications. J Neurotrauma. 2012 May 1;29(7):1364-70. doi: 10.1089/neu.2011.2033. Epub 2012 Feb 22. PMID 22150061
- [Background] Baguley IJ, Nicholls JL, Felmingham KL, Crooks J, Gurka JA, Wade LD. Dysautonomia after traumatic brain injury: a forgotten syndrome? J Neurol Neurosurg Psychiatry. 1999 Jul;67(1):39-43. doi: 10.1136/jnnp.67.1.39. PMID 10369820
- [Background] Baguley IJ, Heriseanu RE, Cameron ID, Nott MT, Slewa-Younan S. A critical review of the pathophysiology of dysautonomia following traumatic brain injury. Neurocrit Care. 2008;8(2):293-300. doi: 10.1007/s12028-007-9021-3. PMID 17968518
- [Background] Mehta NM, Bechard LJ, Leavitt K, Duggan C. Severe weight loss and hypermetabolic paroxysmal dysautonomia following hypoxic ischemic brain injury: the role of indirect calorimetry in the intensive care unit. JPEN J Parenter Enteral Nutr. 2008 May-Jun;32(3):281-4. doi: 10.1177/0148607108316196. PMID 18443140
- [Background] Rabinstein AA, Benarroch EE. Treatment of paroxysmal sympathetic hyperactivity. Curr Treat Options Neurol. 2008 Mar;10(2):151-7. doi: 10.1007/s11940-008-0016-y. PMID 18334137
- [Background] Baguley IJ, Heriseanu RE, Felmingham KL, Cameron ID. Dysautonomia and heart rate variability following severe traumatic brain injury. Brain Inj. 2006 Apr;20(4):437-44. doi: 10.1080/02699050600664715. PMID 16716989
- [Background] Phillips SS, Mueller CM, Nogueira RG, Khalifa YM. A Systematic Review Assessing the Current State of Automated Pupillometry in the NeuroICU. Neurocrit Care. 2019 Aug;31(1):142-161. doi: 10.1007/s12028-018-0645-2. PMID 30484008
- [Background] Miranda A, Taca A. Neuromodulation with percutaneous electrical nerve field stimulation is associated with reduction in signs and symptoms of opioid withdrawal: a multisite, retrospective assessment. Am J Drug Alcohol Abuse. 2018;44(1):56-63. doi: 10.1080/00952990.2017.1295459. Epub 2017 Mar 16. PMID 28301217
- [Background] Mahadi KM, Lall VK, Deuchars SA, Deuchars J. Cardiovascular autonomic effects of transcutaneous auricular nerve stimulation via the tragus in the rat involve spinal cervical sensory afferent pathways. Brain Stimul. 2019 Sep-Oct;12(5):1151-1158. doi: 10.1016/j.brs.2019.05.002. Epub 2019 May 6. PMID 31129152
- [Result] Baguley IJ, Perkes IE, Fernandez-Ortega JF, Rabinstein AA, Dolce G, Hendricks HT; Consensus Working Group. Paroxysmal sympathetic hyperactivity after acquired brain injury: consensus on conceptual definition, nomenclature, and diagnostic criteria. J Neurotrauma. 2014 Sep 1;31(17):1515-20. doi: 10.1089/neu.2013.3301. Epub 2014 Jul 28. PMID 24731076
- [Result] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Result] Kim SW, Jeon HR, Kim JY, Kim Y. Heart Rate Variability Among Children With Acquired Brain Injury. Ann Rehabil Med. 2017 Dec;41(6):951-960. doi: 10.5535/arm.2017.41.6.951. Epub 2017 Dec 28. PMID 29354571
- [Result] Venkata Sivakumar A, Kalburgi-Narayana M, Kuppusamy M, Ramaswamy P, Bachali S. Computerized dynamic pupillometry as a screening tool for evaluation of autonomic activity. Neurophysiol Clin. 2020 Oct;50(5):321-329. doi: 10.1016/j.neucli.2020.09.004. Epub 2020 Oct 11. PMID 33051091
- [Result] Pozzi M, Locatelli F, Galbiati S, Radice S, Clementi E, Strazzer S. Clinical scales for paroxysmal sympathetic hyperactivity in pediatric patients. J Neurotrauma. 2014 Nov 15;31(22):1897-8. doi: 10.1089/neu.2014.3540. Epub 2014 Sep 26. No abstract available. PMID 24964056